CLINICAL TRIAL: NCT01196559
Title: A Phase II Study of Vinorelbine and Gemcitabine Combination In Platinum Resistant Recurrent Epithelial Ovarian/Fallopian Tube/ Primary Peritoneal Carcinoma.
Brief Title: Vinorelbine and Gemcitabine Combination In Platinum Resistant Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Sook Hee Hong, Division of Medical Oncology, Multidisciplinary team of Gynecologic cancer, Seoul St. Mary's hospital, The Catholic University of Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG GY10-10
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Vinorelbine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinorelbine and Gemcitabine (Experimental): Vinorelbine 25 ㎎/㎡ and Gemcibine1000㎎/㎡ D1, D8 every 3weeks
  Interventions: Drug: Vinorelbine and Gemcitabine

INTERVENTIONS:
Drug: Vinorelbine and Gemcitabine — Gmcitabine 1000㎎/㎡ mix in normal saline 100ml iv for 30min andVinorelbine 25㎎/㎡ mix in normal saline 50 ml iv for 5-10min on D1 and 8 every 21 days cycle
  Other Names: Gemcibine and Navelbine

SUMMARY:
The purpose of this study is to evaluate the objective response rate and safety in platinum-resistant epithelial ovarian/fallopian tube/primary peritoneal cancer patients treated with vinorelbine and gemcitabine combination chemotherapy.

DETAILED DESCRIPTION:
Other objectives of this study are to evaluate Progression-free survival and measure CA-125 response rate.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign an approved informed consent form (ICF)
* Histologically or cytologically confirmed epithelial ovarian/fallopian tube/primary peritoneal carcinoma
* Patients had to have received a front-line, platinum/taxane based chemotherapy regimen
* Patients who progressed or whose best response to their most recent platinum-based therapy was less than a partial response will be classified as having platinum-refractory/resistant ovarian cancer or progressed within six months of completing the most recent platinum-based chemotherapy
* Participants must have received prior platinum-based chemotherapy for management of primary disease but must not have received more than 3 prior systemic cytotoxic regimens.
* Patients had to have at least one bidimensionally measurable and/or evaluable (unidimensionally measurable) target lesion in a non-irradiated area and increased Ca 125
* A >= 4 weeks interval between their last chemotherapy regimen and the start of study treatment
* Age 20-75 years old
* Performance status (WHO) 0-2
* Life expectancy of at least three months
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9 gr/mm^3)
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2 mg/dl)

Exclusion Criteria:

* prior therapy with vinorelbine or gemcitabine
* treatment with > 2 cytotoxic regimens (including primary platinum and taxane chemotherapy)
* Serious comorbidities (as determined by the investigator) such as, but not limited to, active congestive heart failure, recent myocardial infarction or active infection.
* Concurrent malignancy requiring therapy (excluding non-invasive carcinoma or carcinoma in situ).
* Symptomatic central nervous system (CNS) metastasis.
* Uncontrolled intestinal obstruction
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy that is considered to be investigational
* Pregnant or nursing.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete response and partial response) | 16 weeks
  radiologically assessed response every two cycles, according to RECIST ver 1.1 criteria and serologically assessed CA 125 response every two cycles, according to Rustin's criteria

SECONDARY OUTCOMES:
Progression Free Survival | 6months
  fom the date of enrollment until the date of confimed progressive disease or death
overall survival | 1year
  from the date of enrollment to death any cause
Frequency and severity of adverse effects | every cycle , from enrollment until death
  assesed by the NCI-CTCAE ver 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ho Byun, Professor, Principal Investigator — Incheon St.Mary;s hospital, Catholic University of Korea; Sook Hee Hong, AP, Principal Investigator — Seoul St.Mary's hospital, Catholic University of Korea
Locations (4):
- South Korea (4):
  - Gyeonsang National University Hospital, Jinju
  - Seoul St. Mary's hospital, Seoul
  - Seoul St Mary's hospital, Seoul
  - Severance hospital, Seoul

REFERENCES:
- [Derived] Hong SH, Lee S, Kim HG, Lee HJ, Jung KH, Lee SC, Lee NR, Yun J, Woo IS, Park KH, Kim KH, Kim HY, Rha SY, Byun JH. Phase II study of gemcitabine and vinorelbine as second- or third-line therapy in patients with primary refractory or platinum-resistant recurrent ovarian and primary peritoneal cancer by the Korean Cancer Study Group (KCSG)_KCSG GY10-10. Gynecol Oncol. 2015 Feb;136(2):212-7. doi: 10.1016/j.ygyno.2014.11.017. Epub 2014 Nov 22. PMID 25462205